CLINICAL TRIAL: NCT03899883
Title: ULTRA-T2D Study: Uric Acid Lowering Trial in Youth Onset T2D
Brief Title: Uric Acid Lowering Trial in Youth Onset T2D
Acronym: ULTRA-T2D
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-1700
Record Dates: First submitted 2019-03-28; First posted 2019-04-02 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Diabetic Kidney Disease; Hyperuricemia; Diabetes; Diabetes Mellitus, Type 2; Type2 Diabetes; Type 2 Diabetes Mellitus; Diabetic Nephropathies; Diabetes Complications
MeSH Terms: conditions — Diabetic Nephropathies; Hyperuricemia; Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Complications | interventions — Pegloticase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pegloticase (Experimental): Single administration of pegloticase (8 mg IV in 250 mL 0.9% normal saline)
  Interventions: Drug: Pegloticase 8 MG/ML [Krystexxa]

INTERVENTIONS:
Drug: Pegloticase 8 MG/ML [Krystexxa] — One time dosing of pegloticase will be administered. Participants will receive an infusion of pegloticase over two hours in the outpatient clinical and translational research center (CTRC) at Children's Hospital Colorado, and will be monitored after infusion.

SUMMARY:
Adolescents and young adults with youth-onset type 2 diabetes (T2D) are disproportionally impacted by hyperuricemia compared to non-diabetic peers and youth with type 1 diabetes (T1D). In fact, 50% of males with youth-onset T2D have serum uric acid (SUA) greater than 6.8 mg/dl. The investigators also recently demonstrated that higher SUA conferred greater odds of developing hypertension and diabetic kidney disease (DKD) in youth with T2D over 7 years follow-up. Elevated SUA is thought to lead to cardiovascular disease (CVD) and DKD by inflammation, mitochondrial dysfunction and deleterious effects on nephron mass. While there are studies demonstrating beneficial effects of uric acid (UA) lowering on vascular health in the general population, there are no studies in youth-onset T2D. Youth-onset T2D carries a greater risk of DKD and CVD compared to adult-onset T2D and T1D.

Accordingly, a clinical trial evaluating UA lowering therapies is needed in youth-onset T2D. Krystexxa (pegloticase), a uricase, effectively lowers SUA and therefore holds promise as a novel therapy to impede the development of CVD and DKD in youth-onset T2D. This proposal describes a pilot and feasibility trial evaluating the effect of UA lowering by pegloticase on markers of CVD and DKD in ten (n=10) youth aged 18-25 with youth-onset T2D (diagnosed <21 years of age) over 7 days. The overarching hypothesis is that pegloticase improves marker of cardiorenal health by lowering UA.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Ages 18-25
* Youth-onset T2D (diagnosis <21 years)
* serum uric acid ≥ 5 mg/dl

Exclusion Criteria:

* Glucose-6-phosphate (G6P) deficiency
* Allergies to seafood or iodine
* MRI contraindications (severe claustrophobia, non-MRI compatible implantable devices, weight ≥ 450 lbs)
* HbA1C ≥ 12%
* Recent (1 month prior) diagnosis of diabetic ketoacidosis (DKA) or hyperosmolar hyperglycemia
* Congestive heart failure
* History of multiple and/or severe allergies or anaphylactic reactions
* Uric acid lowering medications (ie: allopurinol, febuxostat)
* Pegvisomant, pegvaliase, peginterferon alfa 2b, peginterferon alfa 2a, pegfilgrastim, pegaspargase, pegaptanib, pegademase and certolizumab pegol
* Participation in another investigational study within 2 weeks prior to study

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 10 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Markers | 5 min
  Measured by Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP), Mean Arterial Pressure (MAP)
Pulse Wave Velocity (PWV) | 2 hours (x2 study visits)
  Measured by Aortic MRI renal MRI (4D Flow)
Wall Shear Stress (WSS) | 2 hours (x2 study visits)
  Measured by Aortic MRI renal MRI (4D Flow)
Renal Blood Flow | 1 hour (x2 study visits)
  Measured by 4D Flow renal MRI
Glomerular Filtration Rate | 4 hours (x2 study visits)
  Measured by Iohexol Clearance in Plasma
Albumin Excretion Rate (AER) | 4 hours (x2 study visits)
  Measured by albumin and creatinine concentrations in urine

SECONDARY OUTCOMES:
Calculated parameters of intrarenal hemodynamic function | 1 hour
  Measured by using existing renal hemodynamic calculations
Change in serum uric acid (sUA) | 1 hour
  Measured by baseline sUA compared to sUA one week later

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided